CLINICAL TRIAL: NCT02594527
Title: The Southampton Mobility Volunteer Programme to Increase Physical Activity Levels of Older Inpatients: A Feasibility Study
Brief Title: Southampton Mobility Volunteer Programme
Acronym: SoMoVe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RHM MED1297
Record Dates: First submitted 2015-10-19; First posted 2015-11-03 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Physical Activity
Keywords: Older people; Physical activity; Hospital
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteer-led physical activity sessions (Experimental): Patient will receive volunteer-led physical activity sessions twice a day during admission.
  Interventions: Other: Volunteer-led physical activity session

INTERVENTIONS:
Other: Volunteer-led physical activity session — Participants will be encouraged by volunteers to walk or perform chair-based exercises during their stay in hospital

SUMMARY:
Physical activity levels of hospitalised older inpatients is low and this results in many adverse health outcomes. Studies have shown that interventions designed to promote increased physical activity of older inpatients using paid staff have shown improvement in physical function of older inpatients, resulting in shorter hospital stay and reduced admissions to nursing home. This study aims to assess the feasibility and acceptability of using trained volunteers to increase physical activity of older people in hospital. Volunteers will be recruited and trained to encourage older inpatients to mobilise or perform chair-based exercises. Patients will be encouraged to walk or exercise with the volunteers twice a day during their hospital stay. Quantitative analysis will be conducted on the outcome measures. Patients, volunteers and staff members will also be interviewed to assess the acceptability of the intervention. This feasibility study will help inform a future controlled trial.

DETAILED DESCRIPTION:
Background: Previous research has shown that low mobility among older people in hospital is associated with poor health outcomes including worsening physical function and increasing dependence in activities of daily living. There is evidence that the implementation by hospital staff of a mobility or exercise programme for older people in the acute care setting is feasible with promising outcomes including improvement in physical function, shorter hospital stay and reduced nursing home admissions. However employing additional therapy or nursing staff is costly and there are well-recognised shortages of suitable applicants to recruit to these posts. Many National Health Service trusts have an established volunteer workforce and in Southampton trained volunteers have successfully assisted older inpatients at mealtimes.

Objective: This study aims to assess the feasibility and acceptability of using trained volunteers to increase physical activity levels of older people in hospital.

Methods and design: The first part of this feasibility study is the development with the therapy team of a training programme, based on existing literature and best practice, to ensure competency of volunteers in mobilising patients and encouraging physical exercise. The study will be conducted on 2 wards (1 male 1 female) within the Medicine for Older People department. Eligible patients will be encouraged by volunteers to mobilise or perform chair-based exercises, depending on their mobility status, at least twice a day for about 15 minutes each session. The recruitment and retention rates of volunteers will be analysed as will the physical activity interventions they were able to effect. The recruitment of patients, their physical activity and adherence to the intervention will be studied. Qualitative interviews and focus groups will be conducted to explore the views and experiences of the patients, volunteers and health care professionals involved in this study. Participants will be characterised including the measurement of physical activity levels using a StepWatch Activity Monitor and GENEActiv accelerometer. This feasibility study is not powered to show a statistical difference in the outcome measures but data from this study will determine the sample size for future controlled trials.

Discussion: Results from this study will provide valuable information regarding the use of trained volunteers to promote physical activity among older inpatients and the practicalities of implementing the intervention throughout the whole department.

ELIGIBILITY:
Inclusion Criteria:

* deemed appropriate by the medical team and therapists to receive a physical activity intervention by trained volunteers and able to mobilise with or without a walking aid.

Exclusion Criteria:

* patients normally resident in a nursing home, or who were immobile prior to admission;
* patients who are in a side room for infection control reasons;
* palliative care patients;
* patients deemed inappropriate for the physical activity intervention by the medical or therapy teams.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of using trained volunteers to promote increased physical activity among hospitalised older people | 2 year
  Number of volunteers recruited

SECONDARY OUTCOMES:
Acceptability of using trained volunteers to promote increased physical activity among hospitalised older people | 2 years
  Established through interviews and focus groups among patients, volunteers and healthcare staff members.
StepWatch Activity Monitor | 2 years
  Mean step count
GENEActiv accelerometer | 2 years
  Mean acceleration in milligravity
Elderly Mobility Scale | 2 years
Barthel Index | 2 years
Timed Up and Go test | 2 years
Mini-mental state examination | 2 years
Geriatric Depression Score | 2 years
Gait speed | 2 years
Euro-Qol | 2 years
  Measure of quality of life
Length of hospital stay | 2 years
Discharge destination | 2 years
Incidence of thrombotic events | 2 years
Incidence of pressure ulcer | 2 years
Short Form-36 General Health | 2 years
Feasibility assessed by number of volunteers trained | 2 years
Feasibility study assessed by number of volunteers retained | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lim, BM, Principal Investigator — University of Southampton
Locations (2):
- United Kingdom (2):
  - Academic Geriatric Medicine, University of Southampton, Southampton, Hampshire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lim S, Ibrahim K, Dodds R, Purkis A, Baxter M, Rogers A, Sayer AA, Roberts HC. Physical activity in hospitalised older people: the feasibility and acceptability of a volunteer-led mobility intervention in the SoMoVe study. Age Ageing. 2020 Feb 27;49(2):283-291. doi: 10.1093/ageing/afz114. PMID 31566671